CLINICAL TRIAL: NCT04638335
Title: Study to Determine the Proportion of Travelers Over the Age of 60 Years and Travelers Having Lived in a Tropical Country for More Than 5 Years With Anti-HAV Antibodies
Brief Title: What is the Anti-HAV Seroprevalence of Travelers >60 Years or Having Lived in a Tropical Country for >5 Years
Acronym: AHAV
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, Principal Investigator, University of Lausanne Hospitals
Other Study IDs: AHAV-UNIL
Record Dates: First submitted 2020-10-25; First posted 2020-11-20 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- travelers over the age of 60: blood sample taken to test the presence of Anti-HAV antibodies
  Interventions: Biological: Blood test
- travelers having lived in a tropical country for more than 5 years: blood sample taken to test the presence of Anti-HAV antibodies
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — blood test for Anti-HAV antibodies

SUMMARY:
Study to determine the proportion of travelers over the age of 60 years and travelers having lived in a tropical country for more than 5 years with anti-HAV antibodies. This will be done through a blood test. The investigators will then proceed with a short statistical analysis.

DETAILED DESCRIPTION:
Introduction:

Hepatitis A is an infection which is found internationally but mainly in areas where hygiene standards aren't high, as it is transmitted via the fecal-oral route. It is found mainly in Asia, Africa and South America. In these areas, it is mainly children who are infected. The seroprevalence rate reaches close to 100% at 5 years of age in some of these areas. To prevent transmission, following the hygiene recommendations and getting vaccinated are important.

In Switzerland, an average of 60 cases are recorded yearly. These cases are mainly brought in from travelers in countries where hepatitis A is prevalent. Despite this, the prevalence of hepatitis A in Switzerland has diminished over the years. A 1990 study done in Switzerland that measured seroprevalence in different age groups, concluded that it was useful to do a pre-immunisation test in travelers born before 1944 (age 46, now age 75, about a 50% seroprevalence rate), had a history of jaundice or had a prolonged stay (>1 year) in the tropics, subtropics or in Southern Europe. The FOPH (Federal office of public health) has therefore adjusted the vaccination plan to aligne with this conclusion.

Despite the FOPH recommendations, the Expert Committee of Travel Medicine in Switzerland has agreed upon that people who have lived in tropical countries (outside of Europe or North America) for more than 5 years and people who are older than 65 years of age have already developed an immunity against hepatitis A, either through a symptomatic or asymptomatic infection in their infancy. Therefore, they are not vaccinated and their serology isn't tested. The validity of this claim is questionable. Firstly, the level of hygiene has improved in many countries including Switzerland since 1990 when the latest study was done. Secondly, the seroprevalence rate has decreased from 1975 to 2014 in the European Economic Area and European Union. Conversely, the proportion of susceptible people has increased. Thirdly, there is very little circulation of the virus in Switzerland and that has been the case since at least 1988 so there is less of a likelihood that people have gotten infected with the virus. Lastly, In Asia, Latin America, Eastern Europe and the middle East the level of endemicity has decreased over the years due to improved hygienic conditions. Consequently, people that have lived in these countries for 5 years may not have been infected by the virus.

The primary objective is to determine the seroprevalence of anti-HAV in those two groups. The two groups will be analysed separately. If the seroprevalence is >90%, then no vaccination or serology test should be taken. If it is between 50% and 90%, then a serology test should be done first before potentially vaccinating. If it is below 50% then the traveler should be vaccinated.

Method:

This is a cross-sectional mono centric national observational study. The inclusion criteria are people over 60 years old or travelers that have lived in a tropical country for at least 5 years who consult the travel clinic of Unisanté.

The exclusion criteria are if the patient has not consented or is unable to, if they have already been vaccinated against hepatitis A and if they have been injected with immunoglobulines in the past 2 months (half-life of GamaStan: 23 days).

For each participant that has agreed to take part in this project, serum will be drawn. The serum will then be sent to the laboratoire de diagnostic of the CHUV. The results will then be inserted in the patient's case report form. Once about 200 patients (100 for each group) have been collected, a percentage of seroprevalence for each groupe will be determined.

Expected output:

Through this study, the investigators will have a better idea of the seroprevalence in the two groups who are potentially at risk of being infected by Hepatitis A and who are not receiving any preventative measures. The investigators expect that the seroprevalence rate in the two groups will be lower than 90% and therefore the standard of care will need to be changed.

ELIGIBILITY:
Inclusion Criteria:

* people over 60 years old or travelers that have lived in a tropical country for at least 5 years who consult the travel clinic of Unisanté

Exclusion Criteria:

* subjects who have not given their consent,
* are younger than 5 years old,
* are unable to participate for some reason,
* have already been vaccinated against hepatitis A
* have been injected with immunoglobulins in the past 2 months (half-life of GamaStan: 23 days)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: travelers coming for a consultation at the Policlinique de Médecine Tropicale, voyages et vaccinations, Unisanté
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
the percentage of anti-HAV positive tests in the two groups will be calculated | through study completion, an average of 1 year
  In the first groupe, the percentage of travelers over 60 years of age with a positive anti-HAV test will be calculated. In the second groupe, the percentage of travelers having lived for more than 5 years in a tropical country with a positive anti-HAV test will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Serge De vallière, MD,MSc, Principal Investigator — Unisanté
Locations (1):
- Travel Clinic, Department of Ambulatory Care and Community Medicine, University Hospital of Lausanne, Switzerland, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All anonymized data will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be shared within the year of completing the project and will be available for 2 years after first published.